

#### **Informed Consent and HIPAA Authorization Form**

**Study Title:** A Pilot Investigator Initiated Study to Evaluate the Safety, Tolerability and

Efficacy of Elamipretide in the Treatment of Advanced Symptoms of

Friedreich Ataxia (ELViS-FA)

Version Date: March 23, 2023

**Consent Name:** Main Study Consent Form & Study Summary Document

**Principal Investigator:** Dr. David Lynch, MD, PhD Telephone: (215) 590-2242

Emergency Contact: Call the CHOP Operator and

Telephone: (215) 590-1000

ask to speak to the Neurology

Resident on call

You, or your child, may be eligible to take part in a research study. This form gives you important information about the study. It describes the purpose of this research study, and the risks and possible benefits of participating.

In the sections that follow, the word "we" means the study doctor and other research staff. If you are a parent or legal guardian who is giving permission for a child, please note that the word "you" refers to your child.

## Study Overview

You are being asked to take part in this open label research study because you have advanced symptoms of a rare neurological condition called Friedreich ataxia (FRDA).

The purpose of this research study is to find out if an investigational drug called Elamipretide, is safe and effective when used to treat advanced symptoms of FRDA, specifically vision loss and cardiac disease in adults and older children. *Investigational* means that the study drug has not been approved by the US Food and Drug Administration (FDA) and that its use in this study is experimental.

If you agree to take part, your participation will last for 52 weeks (1 year). This research study will involve up to 5 in-person study visits at The Children's Hospital of Philadelphia, as well as study phone calls in between visits. You will receive the study drug, Elamipretide as a daily injection (shot) under the skin (subcutaneous or SC) for 52 weeks. You will be randomized (like the flip of a coin) to either the high dose or low dose group. Once you are randomized, a member of the study team will let you know which group you have been assigned to. After the first 52 weeks, you will have the option to extend for an additional 52 weeks (1 year) if there are signs of clinical improvement, this will involve 1 additional in-person visit at CHOP, with the option to come for an optional in-person visit at Week 68 for an efficacy visit if you wish. Additionally, you will also complete phone calls between study visits.

There are differences between this study and your usual care. As a participant in the research you will:

Receive a study drug; high dose or low dose

· Complete questionnaires and speech testing

CHOP IRB#: IRB 20-018049 Effective Date: 7/17/2024 Expiration Date: 7/16/2025

Page 1 of 19

- Perform various vision tests
- Undergo heart function evaluations
- Have research blood tests at each study visit
- Keep a subject diary

The main risks of the study are from the study drug, Elamipretide. The most frequently reported side effect related to the study drug was reaction to the injection site, such as redness, itching, swelling, and pain. However, it has not been determined if these risks are directly related to the study drug. It should be noted that some side effects may be serious and life-threatening

You may benefit if Elamipretide is effective at stopping or slowing your FRDA symptoms. However, we cannot guarantee that you will receive any direct benefit by participating in this study.

If there is anything in this form you do not understand, please ask questions. Please take your time. You do not have to take part in this study if you do not want to. If you take part, you can leave the study at any time. If you do not choose to take part in this study, you can discuss treatment options with your doctor.

Please see below for additional details about the study.

## What is the current standard of treatment for this disease?

As there is no cure for FRDA, the current standard of care is to treat each symptom individually. For example, your neurologist may recommend that you follow-up with a cardiologist for any heart-related issues, an endocrinologist for any diabetes-related issues, an orthopedic surgeon for scoliosis-related issues, or a physical therapist to help with mobility related issues.

# What is involved in the study?

If you agree to take part in this study, your participation will include receiving either the high dose or low dose of Elamipretide. You will have a 1 in 2 chance, just like the flip of a coin, of receiving either the high dose or low dose. We will then follow you over the course of 52 weeks (1 year). You will be asked to return in-person for study visits at 16 weeks, 36 weeks, and 52 weeks, with study phone calls in between visits. If the study extends into a second year, there will be one additional in-person visit at Week 104 and the option to return at Week 68 in-person if you choose.

Once enrolled, the study drug dose will be determined based on your weight and may be adjusted based on your kidney function. Elamipretide will be administered as a daily subcutaneous (under the skin) injection (shot) that should be performed at the same time each day. The first dose of medication will be administered at your Baseline Visit at CHOP in clinic. You will be required to keep a daily subject diary to report all medication administered and any missed doses.

#### What are the study procedures?

Some of the procedures in this study will be repeated several times. Tests that are part of your regular, routine medical care will continue to be performed. Additional tests may be performed if any of your initial test results are not normal. The study involves the following tests and procedures.

#### **Experimental Procedures:**

Study Drug: You will inject 40-60 mg (high dose) or 20-30 mg (low dose) of Elamipretide by subcutaneous (under the skin) shot daily for the duration of the study. It will need to be injected in your abdomen or thigh. We will train you how to administer the drug. A different area should be used for each dose and you should try to take it at the same time each day. Additional instructional information will be provided to you in the instructions for use document.

#### **Routine Clinical Trial Procedures:**

- Interviews: A team member will take your medical history and demographics. We will also review any medications you are currently taking (prescription and over-the-counter). Throughout the study you will be asked to report if you think that anything bad has happened as a result of the study or if you have had an unwanted side effects from taking the study drug.
- <u>Medical Record Review:</u> We will review your medical records throughout the study to collect information about your medical history (including genetic confirmation of your diagnosis of FRDA), current health, diagnosis, treatments, medications, and results of clinical tests.
- <u>Blood Tests:</u> Blood draws will occur at all in-person study visits in order to see if you can participate in the study, monitor your safety and the effects of the drug, and check your overall health. Depending on the study visit we will collect between 1 and 2 tablespoons of blood at each in-person visit.
  - At the screening visit, your blood will be used to test for HIV and Hepititis B and C. If you are found to have HIV or Hepititis B or C, the results will be shared with you and not with your parent(s). We strongly encourage you to share the results with your parents. Pennsylvania state law requires that all positive HIV test results be reported to the state. If you are found to have HIV or Hepititis B or C, you will not be able to continue participating in the study.
  - The blood draw is a routine procedure with minimal discomfort. We will try not to stick you more than once.
- Randomization: You will be randomly assigned (like the flip of a coin) to one of two groups: the high dose or low dose. You will have a 1 in 2 chance of being assigned to either group.
- <u>Physical Examinations/Vital Signs:</u> Physical exams will be conducted at every inperson visit by the study doctor. The study coordinator will also record your vital signs which will include measurements of weight, height, body mass index, blood pressure, heart rate, breathing rate, and temperature.
- <u>Neurologic Examination:</u> The study doctor will test your movements, speech, balance, and coordination.
- <u>Speech Assessment:</u> You will be asked to complete a series of digital speech assessments. The speech software will collect information about the way you speak. To perform the speech assessment, you will be asked to speak into a microphone which will be recording your voice. This will take about 10 minutes to complete.



- <u>Phone Calls:</u> We will call one week and one month after taking your first dose of study medication to check-in and see how you are doing. We will ask if you have experienced any changes in your health or changes in your medications. Each call will last approximately 15 minutes.
- Questionnaires: You will be asked to complete several questionnaires at each visit. These will ask questions about your daily activities, visual function, and your overall impression of how you are feeling since starting the study drug. Additionally, at the Week 36 (9 month) study visit we will conduct an Exit Interview and ask for your feedback about the study drug, what changes you have noticed, and if you wish to continue in the study. All together, these questionnaires should take about 15 minutes to complete.
- Pregnancy Tests/Urine Sample: For subjects who are female (biological) and have started their periods, a blood sample will be drawn for a pregnancy test at the Screening Visit, unless there is documented evidence confirming they are unable to get pregnant.. The other pregnancy tests will be done at the rest of the visits with a urine sample. If you are found to be pregnant, the results will be shared with you and not with your parent(s). We strongly encourage you to share the results with your parents. If you are found to be pregnant, you will not be able to continue participating in the study.
- Electrocardiograms (ECG): This test measures how fast your heart is beating and whether it is beating normally. If able, you will lie on a bed or table. The cardiology technician will clean several areas on your stomach, chest, rib cage, and back and then attach several small metal disks (electrodes) to the skin on these areas. It may be necessary to clip some hair so the electrodes can properly stick to the skin. The electrodes are hooked to a machine that will trace your heart activity onto a paper. You will be asked to lie very still and breathe normally during the test. You may be asked to hold your breath at certain times.
- Echocardiogram (Echo): An echo makes pictures of your heart using sound waves to check for problems with heart function. We will move a hand-held ultrasound transducer (a special microphone) around your chest to get pictures of your heart. A small amount of clear gel may be applied to your chest to help the transducer work better.
- Heart Magnetic Resonance Imaging (MRI): A heart MRI is a test that is used to obtain an image of your heart. It takes around 45 minutes to complete. You will lie on a table that will move your body into the center of a large magnet that is open at both ends. Utilizing a combination of a large magnet, radio waves, and a computer, several sets of images of your heart will be taken. During the heart MRI, you will receive a solution through an IV. This solution is called gadolinium, and it improves the quality of the pictures taken of your heart.
- <u>Vision Testing</u>: You will be asked to read various vision charts [low contrast (gray letter on white backgrounds), high contrast (black letters on white backgrounds), and dim light (light letters on dark backgrounds)] to the best of your ability using one eye at a time, as well as both eyes at the same time. On each chart the number of correct letters identified is written down. Additionally, you will be asked to download a Vision App on your personal devide that you will be required to complete at all in-person, as well as phone visits.



Optical Coherence Tomography (OCT): You will be asked to have scans of your retinas (in the backs of your eyes) performed using an optical coherence tomography (OCT) machines. This is painless and similar to having photographs taken of the back of your eyes. You will be required to sit still during the brief scanning procedure (a few seconds) for each eye. The OCT scan takes about 15 minutes altogether.

<u>Subject Diary:</u> You will be given study subject drug diaries throughout the study. You will record the date and time you administer the study drug, as well as if you missed any doses.

#### **Visit Schedule**

The table provides a brief description of the purpose and duration of each study visit.

| Visit | Purpose | Main Procedures | Duration |
|---|---|---|---|
| Pre-Visit Day -60 to 0 | Screening Visit | Informed Consent, Medical History, Review Current Medications, Physical and Neurology Examination, Vital Signs, Questionnaires, Serum Pregnancy Testing (if applicable), Blood Tests, Vision Tests, OCT, Vision App, ECG*, Echo*, Speech Testing If all eligibility criteria is met, you can complete | 5-6 Hours |
| | | the Baseline Visit on the same day as the<br>Screening Visit** | |
| <b>Visit 0</b><br>Day 0 | Baseline Visit<br>(Begin Study Drug) | Confirm Eligibility Criteria, Randomization, Review Changes in Medications, Physical and Neurology Examination, Vital Signs, Urine Pregnancy Testing (if applicable), Blood Tests, Vision Tests, OCT, Vision App, ECG, Heart MRI or Echo***, Speech Testing, Questionnaires, Distribute Study Medication and Subject Diary | 5-6 Hours |
| | | Begin Taking Study Drug Daily | |
| <b>Visit 1</b> Day 7 ± 7 | Week 1 Phone Call | Study team will review any changes in your health or changes to your current medications, Vision App | 15 Minutes |
| <b>Visit 2</b> Day 28 ± 14 | Week 4 Phone Call | Study team will review any changes in your health or changes to your current medications, Vision App | 15 Minutes |
| <b>Visit 3</b> Day 112 ± 14 | Week 16 In-Person<br>Visit | Review Changes in Medications, Physical<br>Examination, Vital Signs, Urine Pregnancy Testing (if<br>applicable), Blood Tests, Vision Testing and<br>Questionnaire, ECG, Speech Testing, Return Study<br>Medication and Subject Diary, Dispense New Study<br>Medication and Subject Diary | 2 Hours |
| <b>Visit 4</b> Day 252 ± 14 | Week 36 In-Person<br>Visit | Review Changes in Medications, Physical and<br>Neurology Examination, Vital Signs, Urine Pregnancy<br>Testing (if applicable), Blood Tests, Vision Test, ECG,<br>Heart MRI or Echo***, Speech Testing, OCT, Vision<br>App, Questionnaires (including the Exit Interview),<br>Return Study Medication and Subject Diary, Dispense<br>New Study Medication and Subject Diary | 5-6 Hours |



| <b>Visit 5</b><br>Day 364 ± 14 | Week 52 In-Person<br>Visit<br>(End of Treatment) | Review Changes in Medications, Physical and Neurology Examination, Vital Signs, Urine Pregnancy Testing (if applicable), Blood Tests, Vision Test, ECG, Speech Testing, OCT, Vision App, Questionnaires, Return Study Medication and Subject Diary End of Study Option to Continue into Extension – All subjects will have the option to continue taking the study drug during the Extension until the drug becomes commercially available or the study is terminated. | 4 Hours |
|---|---|---|---|
| Optional Exten | sion | | |
| <b>Visit 6</b> Day 476 ± 14 | Week 68 In-Person<br>(OPTIONAL)<br><u>or</u> | Review Changes in Medications, Physical and<br>Neurology Examination, Vital Signs, Urine Pregnancy<br>Testing (if applicable), Vision Test, OCT, Vision App,<br>Questionnaires, Distribute and Return Study<br>Medication and Subject Diary | 3 Hours |
| <b>Visit 6</b> Day 476 ± 14 | Week 68 Phone Call | Study team will review any changes in your health or changes to your current medications, Vision App | 15 Minutes |
| <b>Visit 7</b> Day 616 ± 14 | Week 88 Phone Call | Study team will review any changes in your health or changes to your current medications, Vision App | 15 Minutes |
| <b>Visit 8</b><br>Day 728 ± 14 | Week 104 In-Person<br>Visit | Review Changes in Medications, Physical and<br>Neurology Examination, Vital Signs, Urine Pregnancy<br>Testing (if applicable), Blood Tests, Vision Test, ECG,<br>Heart MRI or Echo***, Speech Testing, OCT, Vision<br>App, Questionnaires, Return Study Medication and<br>Subject Diary, Dispense New Study Medication and<br>Subject Diary | 5-6 Hours |
| <b>Visit 9</b> Day 756 ± 14 | Week 108 Follow-Up | Study team will review any changes in your health or changes to your current medications, Vision App | 15 Minutes |

- \* If you had an ECG and/or Echo completed within the last 12 months you will not need to perform these tests at the Screening Visit, unless it showed a clinically relevant abnormality, then the procedure will need to be performed at Screening.
- \*\* You will not need to repeat any overlapping study procedures at the Baseline Visit if both the Screening and Baseline Visit are completed on the same day
- \*\*\* Echo's will be offered as an alternative for subjects who are not cardiac MRI compatible, as well as for scheduling conflicts when the cardiac MRI is not available.

# What will be done with my data and specimens during this study?

During the study, we will collect data, as well as blood, and urine samples from you. By agreeing to participate in the study, you agree to give these samples to CHOP for research purposes. As part of this study, if you complete an echocardiogram we will share copies of your de-identified images with the Penn CHPS Echo Team for analysis.

#### Will I receive any results from the tests done as part of this study?

Results that could be important for your clinical care will be shared with you. We will not share other results with you.

## What are the risks of this study?

Taking part in a research study involves inconveniences and risks. The main risks of taking part in this study are discussed below.

## Risks Associated with Study Drug (Elamipretide):

Data from 28 clinical trials have been completed with over 500 human subjects including healthy subjects, as well as patients with various mitochondrial, cardiovascular, renal, visual, and skeletal conditions. The doses used in these studies ranged from 2 mg to 400 mg three times a day.

Injection site reactions were reported in the majority of subjects receiving Elamipretide by SC injection in any study. The most common side effects from injection site reactions included mild redness, swelling, pain, and itching. Generally, the injection site reactions resolved within 4 hours of drug administration. In most studies, the tolerability of the injection site reaction was not problematic and did not require treatment, however some were treated with topical medication to manage the signs and symptoms. Other side effects reported included headaches, dizziness, and infection (such as an upper respiratory tract infection).

There may be other side effects as well that have not been reported or observed yet. An allergic reaction or anaphylaxis to any drug is always a possibility. It is unknown if the study drug Elamipretide will cause an allergic response. If you have a very serious allergic reaction, you may be at risk of death. Some symptoms of allergic reactions are:

- Rash
- Wheezing and Difficulty Breathing
- Dizziness and Fainting
- Swelling around the Mouth, Throat or Eyes
- Fast Pulse
- Sweating

It is important to report any side effects to your doctor. You will be watched after you receive the first dose of Elamipretide for any symptoms that may be an allergy.

Some side effects may be serious and life-threatening.

There may be side effects and discomforts that are not yet known. It is very important that you report any side effect you may experience to your doctor, even if you think it is not related to Elamipretide.

| Adverse Events Related to Elamipretide When Administered Longer Than 8 Days | | |
|---|---|---|
| Common<br>Less then 50 subjects out<br>of 100 | Rare<br>Less then 3 subjects out<br>of 100 | Very Rare<br>Less then 1 subject out<br>of 100 |
| <ul> <li>Injection Site Bruising</li> <li>Injection Site Erythema</li> <li>Injection Site Hemorrhage</li> <li>Injection Site Swelling</li> <li>Injection Site Induration</li> </ul> | <ul><li>Nausea</li><li>Fatigue</li><li>Dizziness</li><li>Headache</li></ul> | <ul> <li>Infected wounds from<br/>injection site reactions</li> <li>Evidence of scar<br/>formation after infected<br/>injection site wound</li> </ul> |

- Injection Site Mass
- Injection Site Pain
- Injection Site Pruritis
- Injection Site Urticaria

# Reproductive Risks Associated with Study Drug (Elamipretide):

The effects of Elamipretide on pregnancy, an unborn baby, and a nursing baby are not well known, there has been one study to date in which exposure during pregnancy occurred with a normal outcome. However, there have been no reports of exposure during lactation, overdoses, or abuse or misuse. In addition, all nonclinical studies (studies conducted using animals or cells rather than human subjects) did not demonstrate any fetal toxicity.

## For Female Subjects:

If you are pregnant or nursing, you will not be allowed to participate in this study. You and your partner will need to take safety measures to prevent pregnancy (such as not having sexual intercourse, or using two medically accepted forms of contraception) for the entire duration of the study, and for at least 30 days after your last dose of study medication.

The study doctor will discuss acceptable forms of contraception with you. If you have questions about how to avoid pregnancy, talk to your doctor or the research team and they will provide you with information on contraceptive choices. You should contact Dr. Lynch at once if you become pregnant during this research study.

#### For Male Subjects:

You should not father a baby during the study and for at least 30 days after your last dose of study medication. You and your partner will need to take safety measures to prevent pregnancy (such as not having sexual intercourse or using an accepted form of contraception) during this time.

The study doctor will discuss acceptable forms of contraception with you. If you have questions about how to prevent pregnancy, talk to your doctor or the research team and they will provide you with information on contraceptive choices.

## Pregnancy Follow-Up:

If you or your partner becomes pregnant during the study, we will ask for permission to follow the pregnancy and collect information on its outcome and the health of your child after birth. If your partner becomes pregnant, we will ask her to sign a separate consent form for this.

#### **Risks Associated with Drug Interactions:**

Some medications may cause unwanted effects when combined with Elamipretide or may make it difficult to tell whether or not the study drug is working. Please tell the study doctor about all of the medications you are taking (including prescription and over the counter drugs, supplements, and vitamins). You should also contact the study doctor before taking any new medications, or stopping or changing any of your current medications. Throughout the study, all possible efforts should be made to maintain stable doses of the medications you take.



The study doctor and staff will discuss with you which medications are allowed and which medications are not allowed during the study. For example, you cannot take systemic, chronic, immunosuppressive drugs. In the event that the FDA approves any new drugs for FRDA during this study, you may not be allowed to enroll in any new clinical trials until after you have stopped taking Elamipretide.

## **Unknown Harms Associated with Study Drug or Other Study Procedures:**

There may be unknown harms or unforeseeable side effects of Elamipretide or the other study procedures. The study doctor and other staff will monitor you closely for any unexpected side effects. We can give you other medicines to make any side effects less serious or to make you feel better.

If you develop any symptoms or conditions during this study, you should notify the study doctor or the emergency contact listed on the cover page of this consent form as soon as possible. If you have an emergency, you should get emergency care. If possible, let the emergency care doctor or nurse know that you are participating in a research study. Also, let the study team know that you had to seek emergency care as soon as possible. For more information about risks and side effects of the study, contact the study doctor, Dr. Lynch.

#### Risks Associated with Neurological and Physical Exams and Pregnancy Testing:

You may experience momentary embarrassment or slight discomfort, however this is unlikely. These procedures are similar to exams and tests that are normally done as part of your routine medical care.

# Risks Associated with the Speech Test, Subject Diaries, Questionnaires, Phone Calls, and Interviews:

You may experience mild fatigue, frustration and/or discomfort or embarrassment while completing these tasks. You can take breaks as needed. You do not have to answer any questions that make you too uncomfortable.

#### Risks of Blood Tests:

Taking blood may cause some pain, bleeding or bruising at the spot where the needle enters your body. Rarely, taking blood may cause fainting or infection.

#### **Risks Associated with ECGs:**

There is a small risk that redness or swelling could develop from the ECG electrodes (pads) that will be placed on the chest.

#### Risks Associated with Echocardiograms:

This procedure is associated with very little discomfort. The gel may feel cold or sticky when first placed on the body. Some people with sensitive skin develop rashes where the wires are taped to the skin. You will feel some mild pressure as the transducer is held against the chest.

#### Risks Associated with Heart MRI:

There are no known risks of physical harm associated with MRI. The sequences are widely used in research worldwide. However, MRI machines produce loud banging noises, which cause some people to become stressed or upset. You may also feel uncomfortable inside the magnet if you do not like to be inside small places or have difficulty lying still. The MRI magnet is always on and attracts certain metal objects.

Any metal objects on or inside of your body may heat up, move, and/or not function properly within the scanning room. Metal objects in the room can fly through the air toward the magnet and hit those nearby. There are many safety measures in place to reduce these risks. The staff will screen all persons and materials entering the scanning room for metal. When the study begins, the door to the room will be closed to minimize the risk of someone accidentally bringing a metal object into the scanner room.

#### Risks Associated with Gadolinium:

Some people may have an allergic reaction to Gadolinium, but this is rare. If this happens, you might experience mild itching, hives, or difficulty breathing which can be a serious life-threatening emergency. If this occurs, it is treatable. Very rarely, gadolinium can cause problems with your kidneys.

#### **Risks Associated with OCT:**

OCT is not a painful procedure. There may, however be some mild discomfort in your eyes.

#### Risks Associated with Breach of Confidentiality:

As with any study involving collection of data, there is the possibility of breach of confidentiality of data. Every precaution will be taken to secure participants' personal information to ensure confidentiality.

At the time of participation, each participant will be assigned a study identification number. This number will be used on data collection forms, blood samples, urine specimens and in the database instead of names and other private information. A separate list will be maintained that will links each participant's name to the study identification number for future reference and communication.

#### Are there any benefits to taking part in this study?

You may benefit by finding some improvement in your FRDA symptoms, such as vision loss or cardiac disease while on the study drug. However, we cannot guarantee or promise that you will receive any direct benefit by participating in this study.

Right now, we do not know if Elamipretide will help treat the advanced symptoms associated with FRDA, however the knowledge gained from this research may help doctors determine the answer to that question. What we learn may help others with FRDA in the future.

#### Do you need to give your consent in order to participate?

If you decide to participate in this study, you must sign this form. A copy will be given to you to keep as a record.

#### What are your responsibilities?

Please consider the study time commitments and responsibilities as a research subject when making your decision about participating in this study. You will need to follow the study doctor's instructions, keep all study appointments and administer the study drug as directed.

**3**H

#### What happens if you decide not to take part in this study?

Participation in this study is voluntary. You do not have to take part in order to receive care at CHOP.

If you decide not to take part or if you change your mind later there will be no penalties or loss of any benefits to which you are otherwise entitled.

## Can you stop your participation in the study early?

You can stop being in the study at any time. You do not have to give a reason.

## Can the study doctor take you out of the study early?

The study doctor may take you off of the study if:

- Your condition worsens.
- The study is stopped.
- The study drug is no longer available.
- You cannot meet all the requirements of the study.
- New information suggests taking part in the study may not be in your best interests.

There may be other reasons that the doctor takes you off of the study.

## What choices do you have other than this study?

There are options for you other than this study including:

- Not participating in this study.
- Receiving care outside this study. Currently, there are no FDA-approved treatments for FRDA.
- You may discuss other options available to you with your doctor.

# What about privacy, authorization for use of Personal Health Information (PHI) and confidentiality?

As part of this research, health information about you will be collected. This will include information from medical records, procedures, interviews and tests that are part of this research. Information related to your medical care at CHOP will go in your medical record. This could include physical exams, imaging studies (heart and vision testing) or blood draws done in the clinical lab. Medical records are available to CHOP staff. Staff will view your records only when required as part of their job. Staff are required to keep your information private. Information that could identify you will not be shared with anyone - unless you provide your written consent, or it is required or allowed by law. Laboratory test results will appear in your medical record with the exception of any blood draws for biomarkers that will be stored for future research, which are performed only for this research study. We will do our best to keep your personal information private and confidential. However, we cannot guarantee absolute confidentiality. Your personal information may be disclosed if required by law.

The results of this study may be shown at meetings and published in journals to inform other doctors and health professionals. We will keep your identity private in any publication or presentation.

3H

Several people and organizations may review or receive your identifiable information. They will need this information to conduct the research, to assure the quality of the data, or to analyze the data or samples. These groups include:

- Members of the research team and other authorized staff at CHOP and Penn
- People from agencies and organizations that perform independent accreditation and/or oversight of research; such as the Department of Health and Human Services, Office for Human Research Protections.
- The Food and Drug Administration (FDA)
- Representatives of Friedreich Ataxia Research Alliance (FARA) and Stealth Biotherapeutics, Inc. who are the study sponsors funding this research
- Your samples will be shared with outside laboratories including Dr. Ian Blair's Lab, who will analyze your samples. Your samples will be labeled with a Study ID number, your initials, and date of sample collection only. The outside laboratories will not know who you are. Private information such as your name, birth date or medical record number will not be shared with them

By law, CHOP is required to protect your health information. The research staff will only allow access to your health information to the groups listed above. By signing this document, you are authorizing CHOP to use and/or release your health information for this research. Some of the organizations listed above may not be required to protect your information under Federal privacy laws. If permitted by law, they may be allowed to share it with others without your permission.

There is no set time for destroying the information that will be collected for this study.

Your permission to use and share the information and data from this study will continue until the research study ends and will not expire. Researchers continue to analyze data for many years and it is not possible to know when they will be completely done.

#### Can you change your mind about the use of personal information?

You may change your mind and withdraw your permission to use and disclose your health information at any time. To take back your permission, it is preferred that you inform the investigator in writing.

Dr. David Lynch
The Children's Hospital of Philadelphia
Division of Neurology/Department of Pediatrics
34<sup>th</sup> Street and Civic Center Blvd.
Philadelphia, PA 19104

In the letter, state that you changed your mind and do not want any more of your health information collected. The personal information that has been collected already will be used if necessary for the research. No new information will be collected. If you withdraw your permission to use your personal health information, you will be withdrawn from the study.



#### **Financial Information**

While you are in this study, the cost of your usual medical care – procedures, medications and doctor visits – will continue to be billed to you or your insurance.

## Will there be any additional costs?

There will be no additional costs to you by taking part in this study. The Study Sponsors are providing financial support and study medication for all experimental producedures completed at The Children's Hospital of Philadelphia for this study.

#### Will you be paid for taking part in this study?

You will be reimbursed up to \$1,000 for travel and hotel expenses per study visit. The reimbursement will be sent to you in the form of checks from The Children's Hospital of Philadelphia within 8 weeks of the study visit. In order to be reimbursed, you will be required to provide documentation of expenses associated with the research visit, including travel, meals, hotel stay, and co-pays. You will also need to complete a Form W-9 or have one on record at CHOP.

You will not receive financial rewards or incentives. There is also no cost to participation in the study. Participants who receive clinical care from the investigator or The Children's Hospital of Philadelphia will be responsible for those charges, as they are separate from the study.

We may share your specimens and data with third parties (other researchers, institutions, or for profit companies). Your specimens and data may be used for commercial profit. You will not receive any financial benefit from the use of your specimens or data.

## Who is funding this research study?

The Friedreich Ataxia Research Alliance (FARA) is providing funding for this study.

In addition, this study is supported by Stealth Biotherapeutics, Inc. Stealth is a drug company that makes the drug being studied in this research project. Stealth is providing the study medication to Children's Hospital for the study at no cost. The results of the study will be reported to both FARA and Stealth. If the study shows that the study drug, Elamipretide may be useful for a new purpose, this could benefit Stealth financially.

Please ask Dr. Lynch if you have any questions about how this study is funded.

# What if you have questions about the study?

If you have questions about this study or how your samples/data are going to be used, call the study doctor, Dr. Lynch at (215) 590-2242. You may also talk to your own doctor if you have questions or concerns.

The Institutional Review Board (IRB) at The Children's Hospital of Philadelphia has reviewed and approved this study. The IRB looks at research studies like these and makes sure research subjects' rights and welfare are protected. If you have questions about your rights and welfare as a subject or if you have a complaint, you can call the Institutional Review Board (IRB) Office at CHOP at (215) 590-2830.

A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify you.

**3**H

At most, the Web site will include a summary of the results. You can search this Web site at any time.

## What happens if you are injured during the study?

If you are hurt or get sick from something that was done as part of this study, doctors at the clinic or hospital can arrange for emergency care. Treatment may be billed to you or your insurer. If your injury is caused by the experimental drug, Stealth may pay for treating the injury. This does not mean that a mistake happened.

The Hospital does not offer financial compensation or payment if you are injured as a result of participating in this research.

If you think you have been injured from taking part in this study, call Dr. Lynch at (215) 590-2242. He can go over things with you, let you know of resources that may be available and give you information on what you need to do.

In case of injury resulting from this study, you will not lose any legal rights by signing this form.

## What will be done with my data and specimens when this study is over?

We may use your data and/or specimens for future research. Sponsors may share the data with researchers/institutions outside of CHOP. This could include for profit companies. We will not ask for your consent before using or sharing them. We will remove identifiers from your data, which means that nobody who works with them for future research will know who you are. Therefore, you will not receive any results or financial benefit from future research done on your data.



#### Optional Consent for Use of Identifiable Data or Specimens for Future Research

As part of the study, we will collect medical information, blood, and urine samples from you. We may wish to use and share this information or samples in a future study about Friedreich ataxia.

Research could occur at CHOP, or at outside institutions, which could include for profit companies. The samples will be given a unique code and will be sent with your age and date of collection but will not include information that can identify you. A master list that can identify you or the blood or urine samples may be kept permanently in a password protected database stored securely on a CHOP network share drive that only study personnel will have access to.

We may not ask for your consent before using or sharing your identifiable specimens or data. You will not receive any results or financial benefit from the future research done on your specimens or data. We may share your identifiable specimens or data with outside researchers who will use them for future research.

If you leave the study, you can ask to have the data collected about you removed or the samples destroyed. You can also ask us to remove information that identifies you from the data or samples. This may not be possible if your samples and data have already been shared.

Please indicate whether you will allow the identifiable data or samples to be used for future research by putting your initials next to one of the following choices:

| (initials | NO, my identifiable (data and/or specimens) may not be used for future<br>research. They may be used for this study only. |
|---|---|
| (initials | ) YES, my identifiable (data and/or specimens) may be used for other future research studies. |



# Consent to Take Part in this Research Study and Authorization to Use and Disclose **Health Information for the Research**

| The research study and consent t | form have been explained to you by: |
|---|---|
| Person Obtaining Consent | Signature of Person Obtaining Consent |
| | Date |
| you agree to take part in this rese<br>to your child's participation. You a<br>information as discussed above. I | cating that you have had your questions answered, earch study and you are legally authorized to consent are also authorizing the use of your/your child's health if you don't agree to the collection, use and sharing of rticipate in this study. <b>NOTE:</b> A foster parent is not a foster child's participation. |
| Name of Subject | |
| Signature of Subject (18 years or older) | Date |
| Name of Authorized Representative (if different than subject) | Relation to Subject: ☐ Parent ☐ Legal Guardian |
| Signature of Authorized Representative | Date |



CHOP IRB#: IRB 20-018049 Effective Date: 7/17/2024 Expiration Date: 7/16/2025

# Child Assent to Take Part in this Research Study

| For children capable of providing assent: | |
|---|---|
| I have explained this study and the procedure terms he/she could understand and that he/sh | |
| Person Obtaining Assent | |
| Signature of Person Obtaining Assent | Date |
| This study has been explained to me a | nd I agree to take part. |
| Signature of Subject (optional) | Date |



#### **STUDY SUMMARY SIGNATURE PAGES**

# For Subjects with Limited English Proficiency

# **Consent to Take Part in this Research Study and Authorization to Disclose Health Information**

| Name of Subject | |
|---|---|
| Name of Authorized Representative (if different than subject) | Relation to Subject: ☐ Parent ☐ Legal Guardian |
| The research study and consent form have guardian. | e been explained to the subject or parent/legal |
| guardian's questions, they have agreed to<br>authorized to consent to their or their child<br>use and share their or their child's health in | at you have answered the subject's or parent's/legal<br>take part in this research study and they are legally<br>'s participation. They have also agreed to let CHOP<br>information as explained above. If they don't agree<br>or their child's health information, they cannot |
| Person Obtaining Consent | Signature of Person Obtaining Consent |
| | _Date: |
| Witness/Interpreter | |
| By signing this form, you are indicating that | at |
| <ul> <li>conveyed by the person obtaining language preferred by and under the subject's questions were into consent were presented in a language.</li> <li>At the conclusion of the consent preferred by and understandable the Summary Document as well</li> </ul> | Document as well as any additional information and consent was presented to the subject in a erstandable to the subject; and the responses of the person obtaining aguage preferred by and understandable to the conference, the subject was asked in a language to the subject if s/he understood the information in as any additional information conveyed by the ding responses to the subject's questions) and |
| Name of Witness/Interpreter | Signature of Witness/Interpreter |
| | Date: |

# Child Assent to Take Part in this Research Study For Subjects with Limited English Proficiency

| For children capable of providing assent: | |
|---|---|
| I have explained this study and the procedure he/she could understand and that he/she free | |
| Person Obtaining Assent | |
| Signature of Person Obtaining Assent | Date |
| <ul> <li>conveyed by the person obtaining language preferred by and underst</li> <li>The subject's questions were interpassent were presented in a langua subject.</li> <li>At the conclusion of the consent copreferred by and understandable to the Summary Document as well as</li> </ul> | ocument as well as any additional information assent was presented to the subject in a tandable to the subject; and preted and the responses of the person obtaining age preferred by and understandable to the onference, the subject was asked in a language of the subject if s/he understood the information in any additional information conveyed by the responses to the subject's questions) and |
| Name of Witness/Interpreter S | Signature of Witness/Interpreter |



Date